CLINICAL TRIAL: NCT03262558
Title: Immunological and Bacteriological Approaches to the Development of Postoperative Mediastinitis With Staphylococcus Aureus
Brief Title: Mediastinitis and Staphylococcus Aureus
Acronym: MEDIASTAPH
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_9886
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Surgery, Cardiac; Infection
Keywords: staphylococcus aureus; nosocomial infection
MeSH Terms: conditions — Infections; Staphylococcal Infections; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with ECC: No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients will undergo standard clinical routine practice in this indication

SUMMARY:
Cardiac surgery with extracorporeal circulation (ECC) yields a deep immune system dysfunction that exposes patients to postoperative infectious complications. Among these, post-operative mediastinitis with Staphylococcus aureus (SA) generates significant morbidity and mortality. Two radically different approaches have been proposed in recent years to reduce the incidence of this complication. A first approach has attempted, without real success, to decrease postoperative immunosuppression. The second, more efficient, consisted of screening and preoperatively treating patients colonized with SA. However, although its incidence has decreased, postoperative mediastinitis remains a terrible nosocomial infection. The authors believe that a thorough analysis of the immunological changes induced by cardiac surgery will initiate active therapeutics to reduce the post-operative immunosuppression phase, thereby decreasing the risk of nosocomial infections. In addition, a study of the interactions between the operated (host) and staphylococcus aureus (pathogenic) immune systems will provide a better understanding of the mechanisms that expose patients to this bacterium.

DETAILED DESCRIPTION:
In particular, changes induced by the ECC will be evaluated on:

* Indoleamine 2,3-dioxygenase activity (IDO)
* Apoptosis of lymphocytes and dendritic cells
* Polymorphonuclear neutrophils (PMNs)
* Myeloid Derived Suppressor Cells (MDSC )

After general anesthesia and arterial catheterization and prior to the start of ECC, blood samples will be taken for flow cytometry studies, for the purification of PMNs and monocytes. The purified PMNs and monocytes will then be used for the measurement of cytokine, phagocytosis and bactericidal production capacities.

The morning following surgery, blood samples will be taken and follow the same process.

ELIGIBILITY:
Inclusion criteria

* Patients over 18 years of age
* Patients who require cardiac surgery (valvular and / or coronary) with extracorporeal circulation.

Non inclusion criteria

* Chronic respiratory diseases,
* Preoperative left ventricular dysfunction (LVEF <50%),
* Immunosuppression (HIV infection, systemic corticosteroid therapy, history of cancer in the year before surgery),
* Persons subject to legal protection (safeguard of justice, curatorship, guardianship),
* Persons deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the aftermath of an ECC for cardiac surgery are investigated to look for the origin of a hypo-reactivity of PMNs and macrophages during exposure to staphylococcus aureus
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-07-04 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-09-29 (Actual)

PRIMARY OUTCOMES:
Variation of plasma IDO activity | Baseline and the morning following surgery
  IDO activity is evaluated by the Kynurenin / Tryptophan ratio before and after ECC.
  Enzymatic activities will be measured by high performance liquid chromatography (HPLC) on pre- and post-operative blood tests

SECONDARY OUTCOMES:
Variation of phagocytosis capacity of PMNs | Baseline and the morning following surgery
  Comparison before and after ECC
Variation of bactericidal capacity of PMNs | Baseline and the morning following surgery
  Comparison before and after ECC
Variation of phagocytosis capacity of macrophages | Baseline and the morning following surgery
  Comparison before and after ECC
Variation of bactericidal capacity of macrophages | Baseline and the morning following surgery
  Comparison before and after ECC
Effect of an inhibitor of IDO on phagocytosis capacities of PMNs | The day following surgery
Effect of an inhibitor of IDO on bactericidal capacities of PMNs | The day following surgery
Effect of an inhibitor of IDO on phagocytosis capacities of macrophages | The day following surgery
Effect of an inhibitor of IDO on bactericidal capacities of macrophages | The day following surgery
Quantification of lymphocytic apoptosis before and after the ECC | Baseline and the morning following surgery
  Quantification of apoptosis by flow cytometry
Quantification of lymphocytic apoptosis in the presence of an inhibitor of IDO | The day following surgery
  Quantification of apoptosis by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TADIE, Md, PhD, Study Director — CHU Rennes
Locations (1):
- Rennes Hospital University, Rennes, France

IPD SHARING:
Plan to Share IPD: No